CLINICAL TRIAL: NCT04454346
Title: Double Foley Catheter For Ripening The Unfavorable Cervix: An Alternative Method
Brief Title: Double Foley Catheter For Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Obut, Medical Doctor, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: 2020/06
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Induction of Labour
Keywords: Double Foley Catheter, Cook balloon, Foley catheter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double Foley Catheter (Experimental): The patients allocated to this arm were randomly and did not differ from the Single Foley Catheter or Cook Balloon arm regard to patients' demographic features and characteristics. The connected FCs were inserted into the cervix using long forceps and advanced to the internal os level. One of the Foley balloons was inflated with 80 ml of saline, and the other FC, now the cervicovaginal balloon, was pulled out with mild traction until the balloon could be visualized and inflated with 20 ml of saline. The vaginal speculum was removed, and the cervicovaginal balloon was inflated further to a total of 80 ml of saline. Both catheters were taped to the inner aspect of the thigh without tension
  Interventions: Device: Double Foley Catheter For Ripening The Unfavorable Cervix
- Single Foley Catheter (Experimental): The patients allocated to this arm were randomly and did not differ from the Double Foley Catheter or Cook Balloon arm regard to patients' demographic features and characteristics. a 16-F FC was inserted into the cervix using long forceps. Then, the balloon was inflated with 80 ml of saline using a standard 20 ml syringe. The catheter was then pulled out until the balloon covered the internal os. The speculum was removed, and the catheter was fixed under slight tension to the inner aspect of the thigh
  Interventions: Device: Double Foley Catheter For Ripening The Unfavorable Cervix
- Cook Balloon (Experimental): The patients allocated to this arm were randomly and did not differ from the Double Foley Catheter or Single Foley Catheter arm regard to patients' demographic features and characteristics. Cook cervical ripening group, the device was applied according to the manufacturer's instructions, and each balloon was inflated with 80 ml saline. The catheter was taped to the inner aspect of the thigh without tension.
  Interventions: Device: Double Foley Catheter For Ripening The Unfavorable Cervix

INTERVENTIONS:
Device: Double Foley Catheter For Ripening The Unfavorable Cervix — New method

SUMMARY:
To compare the efficacy of three mechanical devices for pre-induction of labour cervical ripening: the Single Foley Catheter, Double Foley Catheter (a new handmade device) and Cook cervical ripening balloon.

DETAILED DESCRIPTION:
This prospective study Scheduled included 74 Double Foley Catheter, 74 Single Foley catheter group and 74 Cook cervical ripening catheter group. All pregnant women will be randomly allocated into three groups: the single Foley, Double Foley Catheter or Cook balloon catheter. Removal of the catheters is planned approximately 12 h after insertion if spontaneous expulsion occurred. The main outcome measures include changes in Bishop score, insertion to delivery time, mode of delivery and occurrence of adverse effects.

Double Foley Catheter is a new method for cervical ripening that Two 18-Fr Foley catheters are connected with sterile suture from the hole end and where the balloons borders end. Both catheters are pushed above the internal cervical os the uterus. One of 18-Fr Foley catheter full with 80 mL of normal saline. The other Foley catheter is pulled into the vagina by applying traction and full with 80 mL of normal saline. The cervix between two balloons of Foley catheters exposed to pressure from both sides from the Foley catheter's balloon's similar to Cook balloon.

ELIGIBILITY:
Inclusion Criteria:

* Women with term pregnancy,

Exclusion Criteria:

* Breech presentations, previous cesarean section, Cephalopelvic disproportion, previous uterine scars, estimated fetal weight above 4500

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
vaginal delivery within 24 hours | 24 hours
  the time from applying catheter to delivery
ripening success | 12 hours
  Calculated soon after removal or spontaneous expulsion of catheters above 6 or increasing 2 point above baseline bishop score
pain score | 36 hours
  The pain score during ripening phase which a visual analog scale is completed by the study population to assess the pain score during the entire ripening periods. The pain scores were assessed using the visual analog scale (where 0 = no pain and 10 = worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Obut, M.D, Study Director — Etlik Zubeyde Hanim Woman Health's Care Training and Research Hospital
Locations (1):
- Etlik Zubeyde Hanim Woman's Health Care Training and Research Hospital, Ankara, Turkey (Türkiye)